CLINICAL TRIAL: NCT00164762
Title: Nevirapine Pharmacodynamics and Resistance Among HIV-Infected Mothers in Lilongwe, Malawi
Brief Title: Nevirapine Resistance Study: Nevirapine Resistance Among HIV-Infected Mothers
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kamuzu Central Hospital (Other); University of North Carolina (Other)
Other Study IDs: CDC-NCCDPHP-4535; SIP 26-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections
Keywords: HIV; drug resistance; nevirapine; anti-retroviral drugs; mother-to-child transmission; Treatment Naive; pregnancy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the addition of zidovudine (ZDV) and lamivudine (3TC) at the onset of labor and for up to seven days postpartum to single-dose nevirapine (NVP) is associated with a lower prevalence of NVP-resistant HIV compared to single-dose NVP without ZDV+3TC.

DETAILED DESCRIPTION:
The primary purpose of the Nevirapine Resistance Study is to compare nevirapine (NVP) resistance of HIV at two and six weeks postpartum in women who are participating in two different programs currently ongoing in Lilongwe, Malawi. The first program is through the HIV Infection and Breastfeeding: Interventions for Maternal and Infant Health, also known as the Breastfeeding, Antiretrovirals and Nutrition (BAN) Study, a clinical trial where all enrolled women receive zidovudine (ZDV) and lamivudine (3TC) at the onset of labor and for up to seven days postpartum in addition to single-dose nevirapine (NVP). The second program is the Call to Action (CTA) program sponsored by the Malawi Ministry of Health and Population (MOHP) and UNC Project. The aim of the CTA program is to reduce mother to child transmission (MTCT) of HIV by providing women a single dose NVP to be taken at the onset of labor. Study participants are tested for NVP-resistant HIV at two and six weeks postpartum and the prevalence of NVP-resistant virus is compared among the two groups receiving different peripartum anti-retroviral regimens.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count > 200 cells/μL
* ALT < 2.5 x upper limit of normal (ULN)
* Hemoglobin (Hb) > 7 g/dL
* Age > 18 years, or <18 years and married (considered emancipated minors in Malawi)
* Ability to give informed consent
* Evidence of HIV infection, as documented by 2 positive Enzyme-Linked Immunosorbent Assays (ELISA's); or 1 positive ELISA, and 1 Western blot (WB); or 2 separate concurrent rapid tests. These are the World Health Organization (WHO) acceptable criteria for diagnosing HIV-1 infection in adults.
* Currently pregnant (with a single or multiple fetuses)
* Gestation < 34 weeks
* No serious current complications of pregnancy
* Intention to breastfeed
* Intention to deliver at the institution in which the study is based
* Other than HIV, no active serious infection, such as tuberculosis or other potentially serious illnesses
* No previous use of antiretrovirals including the HIVNET 012 regimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-06; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry L Farr, PhD, Principal Investigator — Centers for Disease Control and Prevention; Denise J Jamieson, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Charles Van der Horst, MD, Principal Investigator — University of North Carolina, Chapel Hill; Peter Kazembe, MB ChB, Principal Investigator — Kamuzu Central Hospital
Locations (1):
- Area 25 Health Center, Lilongwe, Malawi

REFERENCES:
- [Derived] Allen LH, Hampel D, Shahab-Ferdows S, York ER, Adair LS, Flax VL, Tegha G, Chasela CS, Kamwendo D, Jamieson DJ, Bentley ME. Antiretroviral therapy provided to HIV-infected Malawian women in a randomized trial diminishes the positive effects of lipid-based nutrient supplements on breast-milk B vitamins. Am J Clin Nutr. 2015 Dec;102(6):1468-74. doi: 10.3945/ajcn.114.105106. Epub 2015 Nov 4. PMID 26537941
- [Derived] Kayira D, Bentley ME, Wiener J, Mkhomawanthu C, King CC, Chitsulo P, Chigwenembe M, Ellington S, Hosseinipour MC, Kourtis AP, Chasela C, Tembo M, Tohill B, Piwoz EG, Jamieson DJ, van der Horst C, Adair L; BAN Study Team. A lipid-based nutrient supplement mitigates weight loss among HIV-infected women in a factorial randomized trial to prevent mother-to-child transmission during exclusive breastfeeding. Am J Clin Nutr. 2012 Mar;95(3):759-65. doi: 10.3945/ajcn.111.018812. Epub 2012 Jan 18. PMID 22258269
- [Derived] Farr SL, Nelson JA, Ng'ombe TJ, Kourtis AP, Chasela C, Johnson JA, Kashuba AD, Tegha GL, Wiener J, Eron JJ, Banda HN, Mpaso M, Lipscomb J, Matiki C, Fiscus SA, Jamieson DJ, van der Horst C; BAN Study Team. Addition of 7 days of zidovudine plus lamivudine to peripartum single-dose nevirapine effectively reduces nevirapine resistance postpartum in HIV-infected mothers in Malawi. J Acquir Immune Defic Syndr. 2010 Aug;54(5):515-23. doi: 10.1097/qai.0b013e3181e3a70e. PMID 20672451